CLINICAL TRIAL: NCT05748756
Title: The Effect of Bone Marrow Aspirate Concentrate in the Treatment of Mandibular Cystic Defects (Randomized Clinical Trial)
Brief Title: Bone Marrow Aspirate Concentrate in Treating Mandibular Cystic Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BM_22
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Mandible Cyst

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Enucleation and filling by Bone marrow aspirate
- Control group (Active Comparator)
  Interventions: Other: Conventional enucleation only

INTERVENTIONS:
Other: Enucleation and filling by Bone marrow aspirate — The iliac crest is palpated along its widest part forming the iliac tubercle ( 5-6 cm posterior to the anterior superior iliac spine), then a 5 mm incision is made 3-4 cm posterior to the ASIS directly on the crest.
  The needle is advanced between the outer and inner plates of the ileum for a 4-6 cm into the cancellous bone and 10 ml of bone marrow is aspirated.
  Bone marrow aspirate is processed by a dual centrifugation technique.
  Arms: Test group
Other: Conventional enucleation only — patients were treated conventionally by enucleation and plain collagen sponge only.
  Arms: Control group

SUMMARY:
Mandibular cystic defect healing is a complex process. Various methods have been developed to shorten the bone regeneration time and improve its quality. Autogenous grafting is the gold standard for filling cystic defects due to the osteogenesis property provided by the viable cells but is related to donor site morbidity. Allografts and Xenografts are used for the same purpose. However, the increased cost is their main disadvantage. Bone marrow aspirate concentrate is now used to enhance the healing and regeneration process in many areas of the body with no morbidity and low cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from mandibular cystic defect.
* Cystic defect width of 4-8 cm that requires removal under general anesthesia.

Exclusion Criteria:

* Medically compromised patients contradicting operation.
* Previously enucleated lesions.
* Previous surgery, tumor, infection to the pelvis affecting the anterior iliac crest.
* Infected Cysts

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
Change in pain scores | 1st day, 1 week, 4 weeks, 6 weeks
  pain was assessed through a 10-point Visual Analogue Scale (VAS) the scores are categorizied as follows: (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Change in bone density | at baseline, 3 months, 6 months
  An immediate postoperative CBCT was be obtained, followed by another one taken after 3 and 6 months postoperatively. The Region of Interest (ROI) feature was used to estimate the mean bone density in the immediate and 6 months scans. The mean bone density in the 6 months CBCT-scan was compared with the immediate postoperative and the preoperative scans and the mean difference between the scans was calculated.

SECONDARY OUTCOMES:
change in wound dehiscence | 1st day, 1 week, 4 weeks, 6 weeks
  any signs of wound dehiscence were observed

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt